CLINICAL TRIAL: NCT06069882
Title: Cognitive Rehabilitation for People With Mild-to-moderate Dementia: A Single Case Experimental Design Study
Brief Title: Cognitive Rehabilitation for People With Mild-to-moderate Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UGN23NE239
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Dementia
Keywords: Cognitive Rehabilitation; Single Case Experimental Design; Self-efficacy; Goal setting
MeSH Terms: conditions — Dementia | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — Cognitive Rehabilitation is a "person-centred, goal-oriented, problem-solving therapy aimed at managing or reducing functional disability, mitigating excess disability, and maximising engagement and social participation" (Clare et al., 2019, p. 710). For this multiple-baseline SCED, there will be a baseline phase where participants will be assessed on goal attainment without an intervention. This phase will be either 3, 4, 5 weeks long and be determined for the participants using an electronic randomiser programme. Thereafter, facilitators will help participants devise personal rehabilitation plans to achieve one of these goals using evidence-based rehabilitative methods. These methods may include the use of environmental adaptations and prompts, introduction of compensatory strategies, procedural learning of skills, and methods for learning or relearning relevant information. The personal rehabilitation plan is put into practice for 6 weeks during the intervention phase of the study.

SUMMARY:
Cognitive Rehabilitation is an approach that teaches strategies to people with cognitive problems which helps them accomplish tasks which they find challenging. It is found to be helpful for People with Dementia (PwD) who typically are still able to learn new procedures for completing tasks they find difficult. NHS Education for Scotland (NES) have developed a workshop and staff resource that aims to provide health and social care staff in Scotland with the knowledge, skills, and resources to use CR with PwD in a consistent and evidence-based way. The resources developed by the NES are based on the CR in dementia evidence base. However, the usefulness of this programme for Scotland's health services has not been investigated.

The aim of this study is to investigate whether staff assisted use of the CR resources leads to improved goal attainment and self-efficacy for PwD as well as explore the personal experiences of staff, PwD, and their carers of the NES Cognitive Rehabilitation in Dementia intervention, including the impact the intervention may have on participants' confidence in managing their condition.

Six PwD who are seen by Older People's Community Mental Health Teams (OPCMHTs) or the Young Onset Dementia (YOD) service in NHS Greater Glasgow and Clyde (NHSGGC), six nominated persons who act as carers for the PwD, and six clinical team members providing the intervention will have an opportunity to be involved in the study. PwD will develop their own goal related to everyday activities. Their achievement with this goal will be measured many times before and after a CR intervention. The investigators will then investigate if there has been any change in goal success before and after they were given support from staff. The study will also aim to understand the experiences of people participating in CR by conducting interviews with them. The information gathered through the interviews will then be analysed to identify themes in relation to the research aims, such as confidence of PwD in managing their difficulties and facilitators/barriers to participating in the intervention.

The investigators will explore appropriate academic journals with the academic supervisor and submit for publication. The participants will be given the option of receiving a summary sheet of the findings of the study. If successful, the investigators anticipate that the study could encourage greater use of CR interventions to support people with dementia. It is also hoped that insights will offer healthcare providers valuable information when creating services for people with dementia and their carers.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether a Cognitive Rehabilitation (CR) intervention supported by NHS Education for Scotland Cognitive Rehabilitation in Dementia Resources enables people with dementia (PwD) to achieve personally relevant everyday goals, and increases confidence in the ability to manage cognitive difficulties (self-efficacy). Additionally we will explore the personal experiences of staff, PwD, and their carers of the NES Cognitive Rehabilitation in Dementia intervention, including the impact the intervention may have on participants' confidence in managing their condition.

Cognitive Rehabilitation (CR) is an approach that teaches strategies to people with cognitive problems which helps them accomplish tasks which they find challenging. It is found to be helpful for People with Dementia (PwD) who typically are still able to learn new procedures for completing tasks they find difficult. NHS Education for Scotland (NES) have developed a workshop and staff resource that aims to provide health and social care staff in Scotland with the knowledge, skills, and resources to use CR with PwD in a consistent and evidence-based way. The resources developed by the NES are based on the CR in dementia evidence base. However, the usefulness of this programme for Scotland's health services has not been investigated.

Six PwD who are seen by Older People's Community Mental Health Teams (OPCMHTs) or the Young Onset Dementia (YOD) service in NHS Greater Glasgow and Clyde (NHSGGC) will have an opportunity to be involved in the study. The study will use Single Case Experimental Design (SCED) methodology. Participants will develop their own goal related to everyday activities. Their achievement of this goal will be measured between 9-11 times and self-efficacy will be measured six times during the baseline and intervention phases of the study. The combined duration of the baseline and intervention phases is between 9 and 11 weeks. The investigators will then investigate if there has been any change in goal success and self-efficacy before and after they were given support from staff. The study will also aim to understand the experiences of people participating in cognitive rehabilitation for dementia by conducting interviews with them twice, prior to intervention and following the intervention. The information gathered through the interviews will then be analysed to identify themes in relation to the research aims, such as the confidence of people with dementia in managing their difficulties and facilitators/barriers to participating in the intervention.

ELIGIBILITY:
The study will include three participant groups: People with Dementia (PwD), their nominated people and staff participants.

PwD:

Inclusion criteria

* Diagnosis of mild/moderate dementia.
* Currently on the caseload of OPCMHTs or the YOD service in NHSGGC.
* Undergone assessment by OPCMHTs or YOD service and deemed as eligible for CR
* Must have a carer that can act as their nominated person and is able to engage in the intervention and who will also need to provide informed consent.
* If the PwD are taking dementia-specific medication, they need to have been receiving a stable dose for at least one month, with no expectation of change during the trial.
* This study may include those who have a comorbid mental health disorder, brain injury, or other significant neurological disorder, where dementia is still considered by the patient's community mental health team to be the primary presenting difficulty. This is because we often see people who have dementia with comorbid health difficulties.
* They must be proficient in the English language, in order to complete outcome measures.

Exclusion criteria

* A diagnosis of severe/advanced dementia.
* Those who do not have a carer than can act as their nominated person.
* Those who lack the capacity to consent.

Nominated people:

Inclusion criteria

* They must live with the PwD.
* They must be willing to take part in the intervention.
* They must be able to provide informed consent.
* They must be proficient in the English language.

Exclusion criteria • They lack the capacity to consent

Staff participants:

Inclusion criteria

* They must be part of the clinical team.
* They must have health care degree which qualifies them for their post within the clinical team.
* They must be proficient in the English language.
* They must have access to clinical supervision (via a trainee or qualified clinical psychologist) to support their implementation of the NES resources.

Exclusion criteria

• They are not part of the clinical team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-10-17 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment | 9,10, or 11 weeks
  An adapted version of the Goal Attainment Scaling (GAS; Turner-Stokes, 2009) will be used to monitor intervention outcome. On a weekly basis goal achievement status will be recorded using the following GAS categories: (0) at baseline level/no change; (1) partially achieved - some progress from baseline but goal not achieved; (2) goal achieved; (3) more than expected change. In addition, (-1) will refer to deterioration from baseline.
Memory Self-efficacy | 9, 10, or 11 weeks
  The Memory Loss Self-Efficacy Scale (Kurasz et al., 2021) was developed to assess persons with MCI's confidence in performing activities made challenging due to known cognitive deficits. The items on this scale assess self-efficacy for daily activities and managing disease in general, for example "How confident are you that you can do all the things necessary to manage your memory/cognitive difficulties on a regular basis?". Each item is scored on a 10-point scale, from 1 being "Not at all Confident" to 10 being "Totally Confident".

IPD SHARING:
Plan to Share IPD: No
We will not be sharing IPD details to researchers beyond the research team